CLINICAL TRIAL: NCT03193762
Title: Usefulness of a Visual Analogue Scale to Evaluate Anxiety in the Painful Hospitalized Patient
Acronym: EVANX
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Collaborators: Centre Hospitalier de Roubaix (Other); Tourcoing Hospital (Other); Wattrelos hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: OBS-0024; 2017-A00482-51 (Other: ANSM)
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Pain; Anxiety
Keywords: pain; pain management; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders; Agnosia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Painful hospitalized patient: The anxiety of those patients will be measured with an Anxiety VAS
  Interventions: Other: Anxiety VAS

INTERVENTIONS:
Other: Anxiety VAS — Anxiety will be measure with a 10-points visual analogic scale (VAS)

SUMMARY:
Today, there is no simple tool for measuring patient anxiety. The primary purpose of this study is to evaluate the ability of the Visual Analogue Scale (VAS) to measure anxiety in painful hospitalized patients, and to correlate it to STAI-Ya and HAD-7A auto questionnaires.

DETAILED DESCRIPTION:
Pain is one of the major signs, if not the first, which encourages patient to call caregivers. It is a complex and multidimensional sensorial experience. An optimal pain management should consider these different dimensions. If not, the risk is to misidentify pain causes, resulting in therapeutic failures.

Anxiety is one of these dimensions. It's an emotional factor particularly frequent in hospitalized patient.

Pain and hospitalization are both sources of anxiety. Anxiety causes discomfort, hyper vigilance reactions and pain focusing; it can cause avoidance behavior and non-compliance with prescribed medical treatments. Specific care of anxiety can result in a positive impact on hospitalized patient's pains and comfort.

Screening tools for anxiety exist. The STAI-Y is the actual reference scale to measure anxiety. The "Ya" version measures anxiety linked with the reactional state. It's composed of 20 questions and scores of 45 and higher define a significant anxiety (at least moderate). Another tool, the HAD scale, measures anxiety and depression. It has been validated on a population of hospitalized patients. It's composed of 14 questions including 7 about anxiety (HAD-7A). An 11 and higher score defines a significant anxiety (at least moderate). But these tools, theoretically accessible to caregivers, are not often used, especially in hospitalization. The principal reason is their inadequacy to the real conditions in services. Their utilization is too restrictive to hope for an exhaustive diagnosis in routine clinical practice (e.g. the need to have a specific support at disposal or the time to fill in the auto-questionnaires). It would be particularly pertinent to have a faster and easier tool at disposal.

Studies suggest the usefulness of the Visual Analog Scale (VAS) to measure anxiety in pre-operatory or pre-interventional context. This study aims at evaluating VAS' interest in a very frequent situation, the one of painful hospitalized patient. If the VAS demonstrates its capacity to detect and measure anxiety as the validated scales, its utilization could be proposed at the same time as VAS for pain. When pain is assessed by VAS, it'd be easy and simple to evaluate anxiety with the anxiety-VAS, with the same tool, systematically or in anxiety identified situations. Anxious patients who could have specific treatments for anxiety would be better detected and cared for in a general way in accordance with good practice recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Patient hospitalized in a medical or chirurgical service.
* Patient presenting a moderate to acute pain (Pain VAS ≥4)

Exclusion Criteria:

* Patient unable to fill in the auto questionnaire
* Refusal, unwillingness of the patient to participate to the study
* Patients under guardianship, trusteeship and judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Painful hospitalized patient
Sampling Method: Non-Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Correlation between Anxiety VAS and STAI-Ya and HAD-7A scores | at inclusion
  Correlation between Anxiety-VAS and STAI-Ya, HAD-7A scores.

SECONDARY OUTCOMES:
Number of patients presenting anxiety. | at inclusion
  Number of patients presenting significant anxiety according to the different scales used.
Link between anxiety scores and several factors | at inclusion
  The link between the scores at the different anxiety scales and the following factors will be assessed : age, gender, study level, prior hospitalization, antecedent of anxiety-depressive symptoms, treatment, hospitalisation services, reason for hospitalisation, time between hospitalisation and inclusion, painful care, pain origin and pain history
Concordance between STAI-Ya and HAD-7A scales. | at inclusion
  Correlation between STAI-Ya and HAD-7A scores.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ducoulombier, MD, Principal Investigator — Lille Catholic University
Locations (4):
- France (4):
  - Lille Catholic Hospitals, Lille, Nord
  - Roubaix Hospital, Roubaix
  - Tourcoing hospital, Tourcoing
  - Wattrelos hospital, Wattrelos

IPD SHARING:
Plan to Share IPD: No